CLINICAL TRIAL: NCT05218590
Title: For Nasotracheal Intubation With Video Rigid Stylet, Which Nostril is Better? A Randomized Clinical Trial
Brief Title: For Nasotracheal Intubation With Video Rigid Stylet, Which Nostril is Better?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Peking University Hospital of Stomatology (Other)
Responsible Party: Principal Investigator, Yang Xudong, Project leader, Peking University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20220108
Record Dates: First submitted 2022-01-30; First posted 2022-02-01 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Intubation; Video Rigid Stylet
Keywords: Nasotracheal intubation; Nostril; Video rigid laryngoscope

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right nostril group (Active Comparator): Nasal intubation with video rigid stylet was performed through the right nostril.
  Interventions: Device: Video rigid stylet
- Left nostril group (Placebo Comparator): Nasal intubation with video rigid stylet was performed through the left nostril.
  Interventions: Device: Video rigid stylet

INTERVENTIONS:
Device: Video rigid stylet — Nasal intubation was performed using the video rigid stylet.

SUMMARY:
To determine which nostril is more suitable for nasotracheal intubation with video rigid stylet.

DETAILED DESCRIPTION:
Head and neck surgeries usually require nasal intubation, which allows leeway for operative maneuvering in the mouth, pharynx, larynx, and neck. Previous studies have found that the right nostril is more appropriate for nasal intubation using direct laryngoscope or videolaryngoscope. It has been shown that the optical rigid stylet was also an appropriate tool for nasal intubation. However, nasal intubation with rigid optical stylet is technically different from that with laryngoscope. It is unknown whether the choice of nostril could affect the intubation using rigid optical stylet. The main aim is to determine which nostril is more suitable for nasal intubation with video rigid stylet.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. American Society of Anesthesiologists physical status I~II;
3. Scheduled to undergo elective oral and maxillofacial surgery requires nasal intubation;
4. The expected operation time < 3 hours;
5. Extubation in operation room and do not scheduled to preventive tracheotomy;
6. Patients who were able to breathe clearly and equally through both nostrils.

Exclusion Criteria:

1. Patients had history of difficult intubation or presented with an anticipated difficult airway;
2. Patients requiring nasogastric tube insertion;
3. Presence of contraindications of nasal intubation;
4. Due to surgical requirement, intubation must be completed through one nostril;
5. Presence of severe nasal obstruction,deformities of the nasal cavity, or other serious nasal diseases;
6. History of severe epistaxis or epistaxis within a month;
7. Previous history of nasal and/or laryngeal surgery;
8. Previous experience with nasal intubation;
9. History of schizophrenia, Parkinson's disease or profound dementia, or language barrier;
10. Participate in other clinical studies;
11. Refusal to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-16 (Actual)

PRIMARY OUTCOMES:
Total time for intubation | Procedure (From when the device tip entered the nostril to when the tube entered the trachea.)
  The duration from when the device tip entered the nostril to when the tube entered the trachea, as confirmed by capnography.

SECONDARY OUTCOMES:
Total success rate | Procedure (Up to the tube entered the trachea.)
  Total success rate of nasal intubation with video rigid stylet.
First-attempt success | First-attempt of nasal intubation with video rigid stylet.
  First-attempt success of nasal intubation with video rigid stylet.
Times of intubation-attempts | Procedure (From when the device tip entered the nostril to when the tube entered the trachea.)
  Times of intubation-attempts.
The time for device insertion | Procedure (From when the device tip entered the nostril to when it passed through the vocal cord.)
  The duration from when the device tip entered the nostril to when it passed through the vocal cord.
The time for tube insertion | Procedure (From when the tip of the device passed through the vocal cord to when the tube was confirmed inserted into the trachea.)
  The duration from when the tip of the device passed through the vocal cord to when the tube was confirmed inserted into the trachea.
Incidence and severity of epistaxis | Procedure (Up to completion of intubation)
  Incidence and severity of epistaxis

OTHER OUTCOMES:
Intubation related adverse events. | Up to 24 hours after intubation.
  Safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Xudong Yang, MD, PhD, Study Director — Peking University School and Hospital of Stomatology
Locations (1):
- Peking University Hospital of Stomatology, Beijing, China

REFERENCES:
- [Background] Tan YL, Wu ZH, Zhao BJ, Ni YH, Dong YC. For nasotracheal intubation, which nostril results in less epistaxis: right or left?: A systematic review and meta-analysis. Eur J Anaesthesiol. 2021 Nov 1;38(11):1180-1186. doi: 10.1097/EJA.0000000000001462. PMID 34617919
- [Background] Boku A, Hanamoto H, Hirose Y, Kudo C, Morimoto Y, Sugimura M, Niwa H. Which nostril should be used for nasotracheal intubation: the right or left? A randomized clinical trial. J Clin Anesth. 2014 Aug;26(5):390-4. doi: 10.1016/j.jclinane.2014.01.016. Epub 2014 Aug 10. PMID 25113425
- [Background] Cheng T, Wang LK, Wu HY, Yang XD, Zhang X, Jiao L. Shikani Optical Stylet for Awake Nasal Intubation in Patients Undergoing Head and Neck Surgery. Laryngoscope. 2021 Feb;131(2):319-325. doi: 10.1002/lary.28763. Epub 2020 Jun 10. PMID 32521054
- [Derived] Wang LK, Zhang X, Wu HY, Cheng T, Xiong GL, Yang XD. Impact of choice of nostril on nasotracheal intubation when using video rigid stylet: a randomized clinical trial. BMC Anesthesiol. 2022 Nov 24;22(1):360. doi: 10.1186/s12871-022-01910-3. PMID 36424554